CLINICAL TRIAL: NCT03007641
Title: Improving the Approach to and Management of the Older Metastatic Breast Cancer Patient Via a Provider Didactic Intervention
Brief Title: Improving the Approach to and Management of the Older Metastatic Breast Cancer Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-8003
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Provider Didactic Intervention (Experimental): Phase 1 - Providers complete a needs assessment questionnaire.
  Phase 2 - Providers participate in an hour long didactic session, and begin enrolling eligible metastatic breast cancer (MBC) patients. Enrolled MBC patients complete a comprehensive geriatric assessment (CGA). Providers complete a treatment plan questionnaire and a CGA utility questionnaire.
  Phase 3 - Providers are administered a final questionnaire evaluating their overall view of this educational intervention.
  Interventions: Behavioral: Didactic session; Behavioral: Comprehensive Geriatric Assessment

INTERVENTIONS:
Behavioral: Didactic session — This session will include an overview of the approach to and management of older MBC patients through a case-based presentation.
Behavioral: Comprehensive Geriatric Assessment — The Comprehensive Geriatric Assessment (CGA) is a composite of assessment scales evaluating physical, psychological, and social well-being, and is the recommended tool for evaluating an older cancer patient and determining appropriateness of therapy.

SUMMARY:
The purpose of this study is to enhance the care of older metastatic breast cancer (MBC) patients by increasing awareness among oncology providers as to the unique aspects of care required for older patients. The goal of the study is to educate providers on the utility of geriatric assessment in guiding therapy of older metastatic breast cancer patients. The investigators will also assess the feasibility and benefit of incorporating geriatric self-assessments into clinical practice. The study will include three phases.

DETAILED DESCRIPTION:
Older oncology patients pose a significant treatment challenge due to poor chemotherapy tolerance as a result of underlying co-morbidities, lack of social support, and diminished functional reserve. Oncologists are faced with the challenge of differentiating between patients that can and cannot tolerate chemotherapy, and tailoring therapy to the patient's biologic rather than chronologic age.

A significant challenge that surrounds the treatment of the older metastatic breast cancer (MBC) patient in particular, lies in the lack of evidence based clinical data to guide the oncologist in determination of a treatment plan. This is a result of under representation of older patients in clinical trials. Due to these challenges a thorough evaluation of the older patient is recommended prior to initiation of anti-cancer therapy.

The purpose of this research study is to enhance the care of the older MBC patient by increasing awareness among oncology providers as to the unique aspects of care required for older patients. The goal of the study is to educate providers on the utility of geriatric assessment in guiding therapy of older metastatic breast cancer patients. The investigators will also assess the feasibility and benefit of incorporating geriatric self-assessments into clinical practice. The study will include three phases:

1. Needs assessments - to understand the population of older metastatic breast cancer patients seen in routine practice at community centers, and assess their treatment approach.
2. Educational programming about management of older metastatic breast cancer patients, and geriatric assessment of these patients.
3. Active testing of the use of geriatric assessment in clinical practice.

The ultimate goal is to develop an educational curriculum that could be implemented at other community oncology sites beyond the participants on this study. This type of educational intervention can be applied to other disease sites in the future. During the study period we will identify the specific gaps that exist in each practice and develop an educational intervention to match these gaps. Our hope is that all involved practices will benefit from incorporating a geriatric assessment into their practice and will find it feasible to use the tools provided. These data are of high importance to the oncologic community and would be hypothesis-generating for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of metastatic breast cancer (MBC)
* Ongoing active therapy for MBC
* Ability to sign informed consent, and complete a self-assessment evaluation.
* Life expectancy >3 months

Exclusion Criteria:

* No evidence of MBC
* Inability to read and understand English
* Not on active therapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Number of geriatric abnormalities detected | 18 months
  Investigators will test the proportions of patients having at least one abnormality detected by the Comprehensive Geriatric Assessment that was missed in the standard clinical assessment compared to a null-hypothesis rate of 5%.
Percentage of treatment plan changes | 18 months
  Investigators will assess the percentage of physician reported cases whose treatment plan was modified due to responses on the Comprehensive Geriatric Assessment.

SECONDARY OUTCOMES:
Provider perception | 18 months
  Measurement of provider perception of the efficacy and feasibility of the didactic educational session via questionnaire.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - AtlantiCare Cancer Care Institute, Egg Harbor, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Confluence Health, Wenatchee, Washington